CLINICAL TRIAL: NCT00004563
Title: Cyclophosphamide Versus Placebo in Scleroderma Lung Study
Brief Title: Scleroderma Lung Disease
Acronym: SLS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Maureen Mayes, Professor and Elizabeth Bidgood Chair in Rheumatology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 220; U01HL060839 (NIH)
Record Dates: First submitted 2000-02-09; First posted 2000-02-10 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Lung Diseases; Pulmonary Fibrosis; Systemic Scleroderma; Scleroderma, Systemic
Keywords: Lung Diseases; Pulmonary Fibrosis; Systemic Scleroderma; Scleroderma, systemic
MeSH Terms: conditions — Lung Diseases; Pulmonary Fibrosis; Scleroderma, Systemic | interventions — Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cylophosphamide (Experimental): Cyclophosphamide (Cytoxan, Bristol-Myers Squibb) was initiated with a dose of 1 mg per kilogram of body weight per day (to the nearest 25 mg). The doses were increased monthly by one capsule up to 2 mg per kilogram.
  Interventions: Drug: Cyclophosphamide
- Placebo (Placebo Comparator): Matching gel caps at a dose of 25 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide (Cytoxan, Bristol-Myers Squibb) was initiated with a dose of 1 mg per kilogram of body weight per day (to the nearest 25 mg). The doses were increased monthly by one capsule up to 2 mg per kilogram.
  Other Names: Cytoxan (Bristol Myers Squibb)
  Arms: Cylophosphamide
Drug: Placebo — Matching gelcaps 25 mgs
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of cyclophosphamide versus placebo for the prevention and progression of symptomatic pulmonary disease in patients with systemic sclerosis.

DETAILED DESCRIPTION:
BACKGROUND:

Systemic sclerosis is a connective tissue disease of unknown etiology characterized by microvascular injury and excessive fibrosis of the skin and viscera. In the United States, 5,000 to 10,000 new cases are diagnosed annually. Approximately 80 percent of these persons will eventually develop some degree of lung involvement, and restrictive lung disease (interstitial fibrosis) is now the leading cause of morbidity and mortality in systemic sclerosis. An inflammatory alveolitis is thought to be the precursor of interstitial pulmonary fibrosis in systemic sclerosis. An effective treatment for SSc interstitial lung disease has yet to be identified. Cyclophosphamide (CYC) is already being widely used by rheumatologists desperate to do something to halt rapidly declining lung function in SSC patients. Thus, the time is ripe to perform a placebo-controlled trial of CYC in this disease.

Pulmonary scleroderma strikes all races and is most prevalent among women during their child-bearing, child-rearing, and working years. A positive outcome from this trial, demonstrating that oral cyclophosphamide has a beneficial effect on pulmonary fibrosis, would be of great importance by offering a scientific basis for treatment. Similarly, a negative result, demonstrating no benefit from cyclophosphamide therapy, would also be important in avoiding hazardous and expensive therapy that is now being used widely.

DESIGN NARRATIVE:

Multicenter, placebo-controlled, randomized, double-blind. Subjects are recruited at 12 clinical centers and randomized to 2 mg/kg/day of cyclophosphamide or placebo. Follow-up visits for pulmonary assessments occur every three months for two years after treatment. If patients fail the cyclophosphamide treatment, they will be offered azathioprine for the remainder of the 24 month trial. The primary endpoint of the study is change in forced vital capacity at the end of 12 months of treatment. Secondary endpoints include quality of life, activity, and dyspnea indices, and carbon monoxide diffusing capacity. Recruitment ends in December, 2003.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with limited or diffuse systemic scleroderma if they had evidence of active alveolitis on examination of bronchoalveolar-lavage (BAL) fluid (defined as neutrophilia of ≥3 percent, eosinophilia of ≥2 percent, or both)on thoracic high-resolution computed tomography (CT), any ground-glass opacity,
2. Onset of the first symptom of scleroderma other than Raynaud's phenomenon within the previous seven years,
3. An FVC between 45 and 85 percent of the predicted value
4. Grade 2 exertional dyspnea according to the baseline instrument of the Mahler Dyspnea Index (as measured with the use of the magnitude-of-task component).

Exclusion Criteria:

1. A single-breath carbon monoxide diffusing capacity (DlCO) that was less than 30 percent of the predicted value,
2. A history of smoking within the preceding six months, other clinically significant pulmonary abnormalities,
3. Clinically significant pulmonary hypertension requiring drug therapy.
4. Patients taking prednisone at a dose of more than 10 mg per day, those who had previously been treated for more than four weeks with oral cyclophosphamide or had received two or more intravenous doses,
5. Patients who recently received other potentially disease-modifying medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 1999-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Mayes, Principal Investigator — The University of Texas Health Science Center, Houston

REFERENCES:
- [Result] Tashkin DP, Elashoff R, Clements PJ, Goldin J, Roth MD, Furst DE, Arriola E, Silver R, Strange C, Bolster M, Seibold JR, Riley DJ, Hsu VM, Varga J, Schraufnagel DE, Theodore A, Simms R, Wise R, Wigley F, White B, Steen V, Read C, Mayes M, Parsley E, Mubarak K, Connolly MK, Golden J, Olman M, Fessler B, Rothfield N, Metersky M; Scleroderma Lung Study Research Group. Cyclophosphamide versus placebo in scleroderma lung disease. N Engl J Med. 2006 Jun 22;354(25):2655-66. doi: 10.1056/NEJMoa055120. PMID 16790698
- [Derived] Volkmann ER, Wilhalme H, Good S, Kim GHJ, Goldin J, Roth MD, Tashkin DP. A composite endpoint for systemic sclerosis-associated interstitial lung disease: association with mortality in two clinical trial cohorts. Respir Res. 2025 Nov 28;26(1):337. doi: 10.1186/s12931-025-03401-8. PMID 41316297
- [Derived] Khanna D, Clements PJ, Volkmann ER, Wilhalme H, Tseng CH, Furst DE, Roth MD, Distler O, Tashkin DP. Minimal Clinically Important Differences for the Modified Rodnan Skin Score: Results from the Scleroderma Lung Studies (SLS-I and SLS-II). Arthritis Res Ther. 2019 Jan 16;21(1):23. doi: 10.1186/s13075-019-1809-y. PMID 30651141
- [Derived] Kafaja S, Clements PJ, Wilhalme H, Tseng CH, Furst DE, Kim GH, Goldin J, Volkmann ER, Roth MD, Tashkin DP, Khanna D. Reliability and minimal clinically important differences of forced vital capacity: Results from the Scleroderma Lung Studies (SLS-I and SLS-II). Am J Respir Crit Care Med. 2018 Mar 1;197(5):644-652. doi: 10.1164/rccm.201709-1845OC. Epub 2017 Nov 3. PMID 29099620
- [Derived] Namas R, Tashkin DP, Furst DE, Wilhalme H, Tseng CH, Roth MD, Kafaja S, Volkmann E, Clements PJ, Khanna D; Participants in the Scleroderma Lung Study I and members of the Scleroderma Lung Study II Research Group. Efficacy of Mycophenolate Mofetil and Oral Cyclophosphamide on Skin Thickness: Post Hoc Analyses From Two Randomized Placebo-Controlled Trials. Arthritis Care Res (Hoboken). 2018 Mar;70(3):439-444. doi: 10.1002/acr.23282. Epub 2018 Feb 9. PMID 28544580
- [Derived] Kim HJ, Tashkin DP, Gjertson DW, Brown MS, Kleerup E, Chong S, Belperio JA, Roth MD, Abtin F, Elashoff R, Tseng CH, Khanna D, Goldin JG. Transitions to different patterns of interstitial lung disease in scleroderma with and without treatment. Ann Rheum Dis. 2016 Jul;75(7):1367-71. doi: 10.1136/annrheumdis-2015-208929. Epub 2016 Jan 12. PMID 26757749
- [Derived] Khanna D, Nagaraja V, Tseng CH, Abtin F, Suh R, Kim G, Wells A, Furst DE, Clements PJ, Roth MD, Tashkin DP, Goldin J. Predictors of lung function decline in scleroderma-related interstitial lung disease based on high-resolution computed tomography: implications for cohort enrichment in systemic sclerosis-associated interstitial lung disease trials. Arthritis Res Ther. 2015 Dec 23;17:372. doi: 10.1186/s13075-015-0872-2. PMID 26704522
- [Derived] Tashkin DP, Volkmann ER, Tseng CH, Kim HJ, Goldin J, Clements P, Furst D, Khanna D, Kleerup E, Roth MD, Elashoff R. Relationship between quantitative radiographic assessments of interstitial lung disease and physiological and clinical features of systemic sclerosis. Ann Rheum Dis. 2016 Feb;75(2):374-81. doi: 10.1136/annrheumdis-2014-206076. Epub 2014 Dec 1. PMID 25452309
- [Derived] Theodore AC, Tseng CH, Li N, Elashoff RM, Tashkin DP. Correlation of cough with disease activity and treatment with cyclophosphamide in scleroderma interstitial lung disease: findings from the Scleroderma Lung Study. Chest. 2012 Sep;142(3):614-621. doi: 10.1378/chest.11-0801. PMID 22156609
- [Derived] Roth MD, Tseng CH, Clements PJ, Furst DE, Tashkin DP, Goldin JG, Khanna D, Kleerup EC, Li N, Elashoff D, Elashoff RM; Scleroderma Lung Study Research Group. Predicting treatment outcomes and responder subsets in scleroderma-related interstitial lung disease. Arthritis Rheum. 2011 Sep;63(9):2797-808. doi: 10.1002/art.30438. PMID 21547897
- [Derived] Goldin J, Elashoff R, Kim HJ, Yan X, Lynch D, Strollo D, Roth MD, Clements P, Furst DE, Khanna D, Vasunilashorn S, Li G, Tashkin DP. Treatment of scleroderma-interstitial lung disease with cyclophosphamide is associated with less progressive fibrosis on serial thoracic high-resolution CT scan than placebo: findings from the scleroderma lung study. Chest. 2009 Nov;136(5):1333-1340. doi: 10.1378/chest.09-0108. PMID 19892673
- [Derived] Goldin JG, Lynch DA, Strollo DC, Suh RD, Schraufnagel DE, Clements PJ, Elashoff RM, Furst DE, Vasunilashorn S, McNitt-Gray MF, Brown MS, Roth MD, Tashkin DP; Scleroderma Lung Study Research Group. High-resolution CT scan findings in patients with symptomatic scleroderma-related interstitial lung disease. Chest. 2008 Aug;134(2):358-367. doi: 10.1378/chest.07-2444. Epub 2008 Jul 18. PMID 18641099
- [Derived] Strange C, Bolster MB, Roth MD, Silver RM, Theodore A, Goldin J, Clements P, Chung J, Elashoff RM, Suh R, Smith EA, Furst DE, Tashkin DP; Scleroderma Lung Study Research Group. Bronchoalveolar lavage and response to cyclophosphamide in scleroderma interstitial lung disease. Am J Respir Crit Care Med. 2008 Jan 1;177(1):91-8. doi: 10.1164/rccm.200705-655OC. Epub 2007 Sep 27. PMID 17901414
- [Derived] Tashkin DP, Elashoff R, Clements PJ, Roth MD, Furst DE, Silver RM, Goldin J, Arriola E, Strange C, Bolster MB, Seibold JR, Riley DJ, Hsu VM, Varga J, Schraufnagel D, Theodore A, Simms R, Wise R, Wigley F, White B, Steen V, Read C, Mayes M, Parsley E, Mubarak K, Connolly MK, Golden J, Olman M, Fessler B, Rothfield N, Metersky M, Khanna D, Li N, Li G; Scleroderma Lung Study Research Group. Effects of 1-year treatment with cyclophosphamide on outcomes at 2 years in scleroderma lung disease. Am J Respir Crit Care Med. 2007 Nov 15;176(10):1026-34. doi: 10.1164/rccm.200702-326OC. Epub 2007 Aug 23. PMID 17717203

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cylophosphamide | Placebo
Started | 79 | 79
Completed | 54 | 55
Not Completed | 25 | 24
Not completed — Withdrawal by Subject | 20 | 16
Not completed — Lack of Efficacy | 3 | 5
Not completed — Death | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cylophosphamide | Placebo | Total
Number analyzed (Participants) | 79 | 79 | 158
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.2 (1.4) | 47.5 (1.4) | 47.9 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 51 | 111
  Male | 19 | 28 | 47

OUTCOME MEASURES:

1. Primary Outcome: Forced Vital Capacity
Description: The primary end point was the forced vital capacity (FVC, expressed as a percentage of the predicted value) at 12 months, after adjustment for the baseline FVC.
Time Frame: 12 months
Population: The Number of Participants Analyzed is not consistent with the Participant Flow for the following reason: a number of the patients who withdrew, had treatment failure, or died had completed at least the six-month visit--for these patients, a generalized estimating-equation regression model was fitted, and data missing at 12 months were imputed.
Measure: Mean (Standard Error); unit: % of predicted
Arm/Group | Cylophosphamide | Placebo
Number analyzed (Participants) | 73 | 72
% of predicted | 66.6 (1.7) | 65.6 (1.6)

2. Secondary Outcome: Total Lung Capacity
Description: expressed as a percentage of the predicted value
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: % of predicted
Arm/Group | Cylophosphamide | Placebo
Number analyzed (Participants) | 73 | 72
% of predicted | 70.5 (1.8) | 64.7 (1.9)

3. Secondary Outcome: DLCO
Description: diffusing capacity of the lungs for carbon monoxide
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: % of predicted
Arm/Group | Cylophosphamide | Placebo
Number analyzed (Participants) | 73 | 72
% of predicted | 42.8 (1.7) | 44.3 (2.1)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Cylophosphamide | Placebo
Serious Adverse Events (participants affected / at risk) | 5/79 | 5/79
Other Adverse Events (participants affected / at risk) | 20/79 | 4/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cylophosphamide (N=79) | Placebo (N=79)
Leukopenia with pneumonia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia with gastroenteritis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 3 (3)
Pneumonia and Laryngospasm (Renal and urinary disorders) | 3 (3) | 0 (0) — Complicating cystoscopy
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cylophosphamide (N=79) | Placebo (N=79)
Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Hematuria (Renal and urinary disorders) | 9 (9) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 19 (19) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No